CLINICAL TRIAL: NCT01109030
Title: Pioglitazone as an Adjunct for Moderate to Severe Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amirhossein Modabbernia, Dr Amirhossein Modabbernia, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 94976
Record Dates: First submitted 2010-04-17; First posted 2010-04-22 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; pioglitazone; double blind; placebo controlled
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone+Citalopram+Chlordiazepoxide (Active Comparator): Pioglitazone 15 mg Q12h will be given to the patients in active comparator group for 6 weeks. Citalopram 20 mg per day for week one, and then 30 mg/day for 5 consecutive weeks.Chlordiazepoxide 10 mg/day for first three weeks
  Interventions: Drug: Pioglitazone+Citalopram+Chlordiazepoxide
- Placebo+ Citalopram+ Chlordiazepoxide (Placebo Comparator): Placebo 1 Q12h for 6 weeks with the same shape and color as Pioglitazone. Citalopram 20 mg per day for week one, and then 30 mg/day for 5 consecutive weeks.
  Chlordiazepoxide 10 mg each night for first three weeks.
  Interventions: Drug: Placebo+ Citalopram+ Chlordiazepoxide

INTERVENTIONS:
Drug: Pioglitazone+Citalopram+Chlordiazepoxide — Pioglitazone 15 mg every 12 hours for six weeks Citalopram 20 mg per day for week one, and then 30 mg/day for 5 consecutive weeks.
  Chlordiazepoxide 10 mg each night for first three weeks
  Arms: Pioglitazone+Citalopram+Chlordiazepoxide
Drug: Placebo+ Citalopram+ Chlordiazepoxide — Placebo 1 Q12h for 6 weeks with the same shape and color as Pioglitazone. Citalopram 20 mg per day for week one, and then 30 mg/day for 5 consecutive weeks.
  Chlordiazepoxide 10 mg each night for first three weeks
  Arms: Placebo+ Citalopram+ Chlordiazepoxide

SUMMARY:
The purpose of this study is to determine whether Pioglitazone as an adjunct to Citalopram is effective in treatment of moderate to severe depression

DETAILED DESCRIPTION:
Pioglitazone as a Ppar-gamma agonist is an anti diabetic drug. It was also shown that, it has certain anti inflammatory and neuro-protective effects. In recent years it has been proposed that Ppar-gamma agonists may have effects on mood and cognition. In animal studies and in one human case report as well as a pilot study on human subjects these drugs improved symptoms of depression. A randomized controlled and double blind design will provide further evidence for the efficacy of these drugs in major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major depressive disorder based on DSM-IV TR criteria
* Age 18-50
* Hamilton Depression Rating scale >=22
* Signing the informed consent form
* Citalopram be the drug of choice for the patient irrespective of other eligibility criteria

Exclusion Criteria:

* Problems in other Axes
* Pregnancy and lactation
* Serious or life threatening disease
* taking other antidepressant in the recent month or Electroconvulsive shock in the recent two months, and taking other psychotropic agents
* Diabetes controlled with drugs or insulin (patients with only lifestyle interventions will be included), Liver disease, Congestive heart failure Class III and IV
* Metabolic syndrome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Scores of Hamilton Depression Rating Scale (17 items) at the end | week 6
  Hamilton Depression rating scale is a 17-item scale. The questionnaire rates the severity of symptoms observed in depression such as low mood, insomnia, agitation, anxiety and weight loss. The questionnaire is presently one of the most commonly used scales for rating depression in medical research. The primary outcome measure is Scores on Hamilton Depression Rating Scale at the end (week 6)

SECONDARY OUTCOMES:
Number of Adverse events in each group | week 2,4,6
Scores of Hamilton Depression Rating Scale (17 items) | week 0,2,4

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Akhondzadeh, PhD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Department of psychiatry, Roozbeh psychiatric hospital, Tehran University of medical sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Kemp DE, Ismail-Beigi F, Calabrese JR. Antidepressant response associated with pioglitazone: support for an overlapping pathophysiology between major depression and metabolic syndrome. Am J Psychiatry. 2009 May;166(5):619. doi: 10.1176/appi.ajp.2008.08081195. No abstract available. PMID 19411385
- [Background] Rasgon NL, Kenna HA, Williams KE, Powers B, Wroolie T, Schatzberg AF. Rosiglitazone add-on in treatment of depressed patients with insulin resistance: a pilot study. ScientificWorldJournal. 2010 Feb 19;10:321-8. doi: 10.1100/tsw.2010.32. PMID 20191245
- [Background] Rosa AO, Kaster MP, Binfare RW, Morales S, Martin-Aparicio E, Navarro-Rico ML, Martinez A, Medina M, Garcia AG, Lopez MG, Rodrigues AL. Antidepressant-like effect of the novel thiadiazolidinone NP031115 in mice. Prog Neuropsychopharmacol Biol Psychiatry. 2008 Aug 1;32(6):1549-56. doi: 10.1016/j.pnpbp.2008.05.020. Epub 2008 Jun 25. PMID 18579278
- [Background] Eissa Ahmed AA, Al-Rasheed NM, Al-Rasheed NM. Antidepressant-like effects of rosiglitazone, a PPARgamma agonist, in the rat forced swim and mouse tail suspension tests. Behav Pharmacol. 2009 Oct;20(7):635-42. doi: 10.1097/FBP.0b013e328331b9bf. PMID 19745723
- [Result] Sepanjnia K, Modabbernia A, Ashrafi M, Modabbernia MJ, Akhondzadeh S. Pioglitazone adjunctive therapy for moderate-to-severe major depressive disorder: randomized double-blind placebo-controlled trial. Neuropsychopharmacology. 2012 Aug;37(9):2093-100. doi: 10.1038/npp.2012.58. Epub 2012 May 2. PMID 22549115